CLINICAL TRIAL: NCT01740284
Title: A Phase III Trial Evaluating Tolerability of Grazax Treatment in Combination With Antihistamine in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis
Brief Title: A Trial Evaluating Tolerability of Grazax Treatment in Combination With Antihistamine
Acronym: GT-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GT-19
Record Dates: First submitted 2012-11-14; First posted 2012-12-04 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Allergic Rhinoconjunctivitis
MeSH Terms: interventions — Grazax; desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazax + Aerius (Active Comparator): 1 tablet (oral lyophilisate ) on Day 14 and Day 28 of Grazax (Phleum Pratense grass pollen allergen extract) 75.000 SQ-T and 1 tablet (melting tablet)of Aerius (desloratidine) 2.5 mg
  Interventions: Drug: Grazax + Aerius
- Grazax + Placebo (Placebo Comparator): 1 tablet (oral lyophilisate ) on Day 14 and Day 28 of Grazax (Phleum Pratense grass pollen allergen extract) 75.000 SQ-T and 1 tablet (melting tablet)of Aerius (Placebo)
  Interventions: Drug: Grazax + placebo

INTERVENTIONS:
Drug: Grazax + Aerius
  Arms: Grazax + Aerius
Drug: Grazax + placebo
  Arms: Grazax + Placebo

SUMMARY:
Many grass pollen allergic subjects treated with immunotherapy tablets experience treatment related adverse events when initiating treatment.

The majority are local allergic reactions within the mouth and/or throat, and most of these reactions are mild or moderate. It is anticipated that intake of antihistamine before initiation of Grazax treatment would most likely reduce the discomfort associated with initiation of Grazax treatment. So this trial was to investigate if administration of antihistamine prior to initiation of Grazax treatment results in a reduction of subjects reporting local allergic reactions.

DETAILED DESCRIPTION:
Many grass pollen allergic subjects treated with immunotherapy tablets experience treatment related adverse events when initiating treatment. The adverse events are considered consistent with the introduction of allergens in sensitised subjects. The majority are local allergic reactions within the mouth and/or throat. Most of these reactions are mild or moderate in intensity, have an onset almost immediately after taking a tablet, and last from minutes to hours after intake. Appearance of adverse events in relation to tablet intake tends to subside spontaneously within 1 to 7 days. Thus, initiation of treatment with Grazax may be associated with discomfort. It is anticipated that intake of antihistamine before initiation of Grazax treatment would most likely reduce the discomfort associated with initiation of Grazax treatment. Therefore, the rationale for this trial was to investigate if administration of antihistamine prior to initiation of Grazax treatment results in a reduction of subjects reporting local allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age
* Written informed consent obtained before any clinical trial procedures are performed
* A clinical history of grass pollen induced allergic rhinoconjunctivitis of two years or more requiring treatment during the grass pollen season
* Reporting of treatment related allergic AEs (local reactions in mouth and throat) after intake of Grazax at screening (visit 1)
* Positive skin prick test (SPT) response (wheal diameter ≥ 3 mm larger than the negative control with a flare) to Phleum pratense
* Female subjects had to be non-pregnant and non-lactating.
* Subject willing and able to comply with the protocol

Exclusion Criteria:

* Uncontrolled asthma in the past 12 months
* FEV1 < 70% of predicted value (calculated according to ECCS (20))
* A clinical history of symptomatic seasonal allergic rhinitis and/or asthma due to another allergen which might have caused symptoms during the conduct of this trial
* A clinical history of significant symptomatic perennial rhinitis or allergic rhinitis/asthma caused by an allergen to which the subject was regularly exposed
* At randomization, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process (serous otitis media is not an exclusion criterion)
* History of emergency visit or admission for asthma in the previous 12 months
* Use of an investigational drug within 30 days prior to screening
* History of anaphylaxis, including anaphylactic food allergy, insect venom anaphylaxis, exercise anaphylaxis or drug induced anaphylaxis
* History of chronic urticaria within the last year
* History of angioedema
* Any of the following underlying conditions known or suspected to be present:
* Cystic fibrosis, malignancy, insulin-dependent diabetes, malabsorption or malnutrition, renal, or hepatic insufficiency, chronic infection, drug dependency or alcoholism
* Any evidence of disease making implementation of the protocol or interpretation of the protocol results difficult or jeopardising the safety of the subject (e.g. clinically significant cardiovascular, serious immunopathologic, immunodeficiency whether acquired or not, hepatic, neurologic, psychiatric and ongoing long term treatment with tranquilizer or psychoactive drugs, endocrine, or other major systemic disease or malignancies (including auto-immune diseases, tuberculosis and HIV)).
* Immunosuppressive treatment
* History of allergy, hypersensitivity or intolerance to IMPs (except for Phleum pratense) or desloratadine
* Unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the trial, which in the opinion of the investigator will compromise the data
* Being the investigator, trial staff or their immediate families, defined as the investigator's/staff's spouse, parent, child, grandparent, or grandchild or being the 2nd member of a family (living in the same household)
* Use of any prohibited drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate whether intake of antihistamine in connection with Grazax treatment results in a reduction in number of subjects reporting treatment related AEs the first day of Grazax exposure | 28 days following the first dosing

SECONDARY OUTCOMES:
Other safety endpoint | 28 days following first dosing
  Vitals signs measured three times (Day 0, Day 14 and Day 28)
Other safety endpoint | 28 Days following the first dosing
  FEV1 measured three times (Day 0, Day 14 and Day 28)

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für Rhinologie und Allergologie, Wiesbaden, Germany